CLINICAL TRIAL: NCT06229535
Title: The Right to be Forgotten in the AYA Population: Patients' Experience and Perspectives (Diritto All'Oblio)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-21
Record Dates: First submitted 2023-12-12; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Oncologic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer survivors experience a form of social discrimination that is described in numerous areas such as private life, educational and work paths and the achievement of personal goals. Starting from this scenario, more and more national legislative initiatives are emerging to reconcognize the right to be forgotten, defined as the right not to have to report one's, resolved, oncological disease in contact with institutions such as insurance companies, banks or others. The issue of the right to be forgotten is current and new, primarily in the AYA (adolescents and young adults) population. The purpose of this study is to explore and describe the experience of adolescents and young adults affected by previous oncological disease with respect to the issue of the right to be forgotten. In particular, focusing on:

* awareness (knowledge of the issue);
* significance attributed and subjective perception;
* implications/fallouts perceived or experienced on one's present and future history.

DETAILED DESCRIPTION:
Cancer survivors experience a form of social discrimination that is described in numerous areas such as private life, educational and work paths and the achievement of personal goals. Starting from this scenario, more and more national legislative initiatives are emerging to reconcognize the right to be forgotten, defined as the right not to have to report one's, resolved, oncological disease in contact with institutions such as insurance companies, banks or others. The issue of the right to be forgotten is current and new, primarily in the AYA (adolescents and young adults) population. The purpose of this study is to explore and describe the experience of adolescents and young adults affected by previous oncological disease with respect to the issue of the right to be forgotten. In particular, focusing on:

* awareness (knowledge of the issue);
* significance attributed and subjective perception;
* implications/fallouts perceived or experienced on one's present and future history.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis between (or equal to) 15 and 39 years;
* patients not in active phase of treatment;
* at least 5 years elapsed since diagnosis;
* comprehension and written expressive ability of the Italian language.
* subscription informed consent to the study.

Exclusion Criteria: NA

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50-60 subjects afferent to pediatric and adult oncology centers, off therapy for at least 1 year and with at least 5 years since the diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2024-11-16 (Estimated)

PRIMARY OUTCOMES:
Frequency of participants citing words attributable to the topic of awareness in the text with the aim to explore the experience of adolescents and young adults with prior cancer with respect to the issue of the right to be forgotten. | up to 1 year
  Frequency with which words attributable to the topic of awareness are expressed in the text
Frequency of participants citing words attributable to the thematic area that delineate the architecture of the text about meaning and subjective perception of the right to be forgotten. | up to 1 year
  Frequency of participants citing words attributable to the thematic area that delineate the architecture of the text about meaning and subjective perception of the right to be forgotten.
Frequency of participants citing words attributable to implications/implications perceived or experienced on one's present and future history with respect to the issue of the right to be forgotten. | up to 1 year
  Frequency of participants citing words attributable to implications/implications perceived or experienced on one's present and future history with respect to the issue of the right to be forgotten.

SECONDARY OUTCOMES:
Frequency of patients with information that can lead to the recognition of the right to be forgotten primarily in the AYA population | up to 1 year
  Frequency of patients with information that can lead to the recognition of the right to be forgotten primarily in the AYA population measured through indicators that identify this argumentative junction in the text

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Mascarin, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Francesca Bomben, Dr, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (9):
- Italy (9):
  - Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Università degli studi di Milano - Bicocca, Monza
  - Università di Palermo, Palermo
  - IRCCS, Ospedale Bambino Gesù, Roma
  - Ospedale Regina Margherita, Torino